CLINICAL TRIAL: NCT03807921
Title: Randomized Control Study of Anticoagulation With Warfarin Por Patients With Aortic Bioprosthesis vs Aspirin Only
Brief Title: Anticoagulation for Aortic Bioprosthesis (ANTIPRO)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Cirugia Cardiaca, Uruguay (Other)
Collaborators: Universidad de la Republica (Other)
Responsible Party: Principal Investigator, Victor Dayan, Cardiac Surgeon, Instituto Nacional de Cirugia Cardiaca, Uruguay
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANTIPRO
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve Insufficiency; Aortic Valve Regurgitation
Keywords: aortic valve replacement; bioprosthesis; anticoagulation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Disease; Aortic Valve Insufficiency | interventions — Warfarin; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warfarin (Experimental): Warfarin will be started 48-72h after aortic valve replacement. Dose will be 5 mg daily in order to obtain an Internation normal ratio (INR) of 2-3. Warfarin treatment will continue for 3 months.
  Aspirin will be administered 100 mg daily.
  Interventions: Drug: Warfarin; Drug: Aspirin
- Aspirin only (Active Comparator): Aspirin will be started 48-72h after aortic valve replacement. Dose will be 100 mg daily. Patients who undergo coronary artery revascularization will receive 325 mg daily.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Warfarin — Oral anticoagulation
  Other Names: Choice
  Arms: Warfarin
Drug: Aspirin — Antiplatelet treatment
  Other Names: AAS

SUMMARY:
This study evaluates the clinical and hemodynamic outcome in patients after aortic valve replacement. Half of the patients will receive warfarin + aspirin and the other half will receive only aspirin. The investigators will focus mainly on early bioprosthesis degeneration.

DETAILED DESCRIPTION:
Aortic bioprosthesis have the advantage that they do not require life-long anticoagulation. Current guidelines support the use of aspirin (AAS) 100 mg as a class I indication.

Current evidence, mainly derived from transaortic valve implantation (TAVI) patients, have shown that aortic bioprosthesis suffer subclinical thrombosis which may explain the increase in gradient and bioprosthetic degeneration. Anticoagulation in this cases improve leaflet mobility and decrease in gradient. Evidence supporting early anticoagulation in patients with aortic bioprosthesis is not as strong as in the case of mitral bioprosthesis. Nonetheless, current American Heart Association/American College of Cardiology (AHA/ACC) guidelines recommend (IIa) the use of warfarin for at least 3 months after aortic valve replacement.

The aim is to conduct a single blinded (echocardiographist) randomized control study in patients who receive an aortic bioprosthesis. Comparison will be performed between the use of warfarin + aspirin vs aspirin alone. Duration of anticoagulation will be for 3 months and patients follow-up for 1 year. Clinical and echocardiographic evaluation will be performed in every patients. Some patients will undergo Positron Emission Tomography (PET-Scan).

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of aortic valve replacement with porcine bioprosthesis

Exclusion Criteria:

* Concomitant mitral valve replacement
* Previous atrial fibrillation
* Previous use oral anticoagulation
* Contraindication for the use of oral anticoagulation (high risk of bleeding, intolerance, allergy)
* Jehovah witness
* Platelet count below 90,000.
* Liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Transprosthetic aortic gradient | 3 months and 1 year
  Change in Transprosthetic mean gradient
Change in New York Heart Association (NYHA) class | 1 year
  NYHA class

SECONDARY OUTCOMES:
Major bleeding | 3 months and 1 year
  number of patients admitted due to Genitourinary (GU) or Gastrointestinal (GI) bleeding, pericardial tamponade, pleural effusion
Embolic events | 3 months and 1 year
  Number of patients with cerebral and peripheral ischemic events
Prosthetic leak | 3 months and 1 year
  Change in severity of prosthetic and paraprosthetic leakage

CONTACTS AND LOCATIONS:
Overall Officials: Victor Dayan, MD, PhD, Principal Investigator — Instituto Nacional de Cirugia Cardiaca; Diego Freire, MD, Principal Investigator — Centro Cardiovascular Universitario
Locations (2):
- Uruguay (2):
  - Centro Cardiovascular Universitario, Montevideo
  - Instituto Nacional de Cirugia Cardiaca, Montevideo

IPD SHARING:
Plan to Share IPD: Yes
Study protocol.
Supporting Information: Study Protocol, ICF
Time Frame: From January 2019
Access Criteria: Protocol will be shared by email. Investigators interested should send email to the PI who will evaluate the solicitude.